CLINICAL TRIAL: NCT03897985
Title: Measurement of Anaesthesia-depth Trough Narcotrend TM in Patients Undergoing Electro-Convulsion-Therapy (ECT)- Influence of Anaesthesia Depth on Quality of Convulsion - A Non-Intervention Trial
Brief Title: Measurement of Anaesthesia-depth Trough Narcotrend TM in Patients Undergoing Electro-Convulsion-Therapy (ECT)- Influence of Anasthesia Depth on Quality of Convulsion
Acronym: TM TradeMark
Status: Completed | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: Narcotrend-ECT Study
Record Dates: First submitted 2019-03-29; First posted 2019-04-01 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2019-03

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Narcotrend TM — Measurement of anesthesia depth

SUMMARY:
The Electro-Convulsion-Therapy (ECT) is a well accepted treatment option in severe depression. The quality of ECT is evaluated basing on minimal seizure duration (>15sec), the sympathic response and the postictal EEG-suppression.

For the treatment general anaesthesia is needed. On the other hand anaesthesia strongly influences the quality of the seizure. The goal is to find an anaesthesia-depth that is needed for the well-being of the patient and allows a good ECT.

In daily routine the dose of anesthetic agents and the assesment of anesthesia-depth is based on the subjective estimation of the anesthetist and also on ealier interventions.

The aim of the study is to assess any correlation between measured anesthesia-depth using the Narcotrend TM and the Quality of the ECT.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) Physical Satus I-3
* >18 years < 90 years
* Signed informed consent

Exclusion Criteria:

* Refusal of the patient

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient sceduled for elective ECT for the Treatment of severe deppression
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Correlation of anesthesia depth measured by Narcotrend TM and quality of ECT treatment | 1 day

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Austria

REFERENCES:
- [Derived] Gasteiger L, Heil M, Horner E, Andexer J, Kemmler G, Hausmann A, Lederer W. Relationship Between Anesthesia Depth and Quality of Seizures in Patients Undergoing Electroconvulsive Therapy: A Prospective Observational Study. J ECT. 2022 Mar 1;38(1):62-67. doi: 10.1097/YCT.0000000000000792. PMID 34519686